CLINICAL TRIAL: NCT01524471
Title: Per-Oral Endoscopic Myotomy (P.O.E.M.) for Treatment of Primary Esophageal Motility Disorders
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CRE_2010.430
Record Dates: First submitted 2012-02-01; First posted 2012-02-02 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Achalasia
Keywords: Hypertensive LES
MeSH Terms: conditions — Esophageal Achalasia

ARMS (1):
- POEM (Experimental): Endoscopic Myotomy
  Interventions: Procedure: Per Oral Endoscopic Myotomy

INTERVENTIONS:
Procedure: Per Oral Endoscopic Myotomy

SUMMARY:
Spastic esophageal motility disorders induced significant symptoms including dysphagia, retrosternal pain and regurgitation. Per oral endoscopic myotomy (P.O.E.M.) is a novel approach to perform myotomy through the esophagus with long submucosal tunnel. This study aimed to investigate the feasibility and safety of P.O.E.M. and translate the techniques from animal study to clinical practice in human.

ELIGIBILITY:
Inclusion Criteria:

* All patients with age ranged 18 to 80 who had primary esophageal motility disorders will be recruited. The primary motility disorders included: Achalasia, hypertensive LES, Nutcracker esophagus and Diffuse esophageal spasm.

Exclusion Criteria:

* Patients will be excluded from this study with the followings -

  1. Pregnancy
  2. Informed consent not available
  3. Previous history of esophagectomy or mediastinal surgery
  4. Previous history of endoscopic resection for early esophageal cancers, including endoscopic mucosal resection and endoscopic submucosal dissection
  5. End-stage Achalasia with dilated esophagus more than 6cm on Barium swallow Investigations before and after POEM

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Dysphagia score

SECONDARY OUTCOMES:
Improvement in LES pressure
Eckhart score
Operative time
Length of myotomy
Time to resume diet
Morbidities

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Chinese University of Hong Kong, Hong Kong, Hong Kong